CLINICAL TRIAL: NCT06543732
Title: Vital@Work: a Personalized Reintegration Program for Employees with Stress-related Complaints
Brief Title: Vital@Work: Reintegration Program for Employees with Stress-related Complaints
Acronym: Vital@Work
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Health Holland (Other); Trimbos (Unknown)
Responsible Party: Principal Investigator, Trees Juurlink, Senior researcher, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024.0021
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Return to Work; Mental Health
Keywords: Return to work; Stress; Absenteeism
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing intervention group with care as usual group. Randomization is carried out at the individual level stratified by organisation type and whether problems are perceived as work-related or not.
Who Masked: Participant
Masking Description: Due to the PA intervention, it is not possible to blind the researchers and process facilitators. However, workers randomized to the intervention or control group are not aware of the research design. Process facilitators providing the PA are informed about the research design and the outcome of randomization, and they are asked not to communicate the research design to the employees.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eHealth with Participatory Approach if needed (Experimental): Participants receive a personalized eHealth program and if needed, after 6 weeks the Participatory Approach (intervention) next to care as usual from occupational health care.
  Interventions: Other: Return to work program
- Control condition (No Intervention): Participants receive links to existing websites on return to work next to care as usual from occupational health care.

INTERVENTIONS:
Other: Return to work program — The eHealth modules focus on psychoeducation, perceptions of return to work based on a personal plan including problem-solving exercises, relapse prevention, and continuous monitoring. If needed, followed by the participatory approach, a stepwise, collaborative approach to analyse and solve bottlenecks to develop a consensus-based plan for return to work.
  Arms: eHealth with Participatory Approach if needed

SUMMARY:
The objective of this study, Vital@Work reintegration program, is to support sick-listed workers with stress-related complaints in their return to work based on a personalized program. Therefore, the aim of this study is test whether participants supported by a tailored eHealth program, and if needed, additionally supported by a structured and stepwise Participatory Approach (PA) involving the sick-listed worker, their direct supervisor and a neutral party, show a faster and sustainable return to work as compared to participants in the control condition. This program is investigated in four different organizations, which differ in sector, size (small and large organizations), type of organization (private or public) and type of work.

DETAILED DESCRIPTION:
This study evaluates the effectiveness of a program, incorporating diverse components, to improve sustainable return to work, stress-related outcomes and cost effectiveness among sick-listed workers with stress-related complaints compared to usual care. The study design is a randomized controlled trial, including an intervention and control group. Sick-listed workers between 2 - 12 weeks sick, in the intervention group receive a tailored eHealth program based on their questions on a distress screener, if needed followed by the Participatory Approach (PA). Sick-listed workers in the control group receive standard practice and general information about return to work. If sick-listed workers did not return to work after 6 weeks in the eHealth program, the PA starts. The PA is a structured and stepwise procedure that involves the sick-listed worker, their direct supervisor, and a neutral party (either physically present or working in the background) to guide the conversation. This collaborative process aims to identify workplace-related bottlenecks, and subsequently develop a consensus-based return to work plan based on a strong commitment of both the sick listed worker and employer. This study offers two different forms of PA: individual work modifications (guided by a neutral process facilitator) and job coaching (guided by the employer, with the process facilitator providing support in the background). If sick-listed workers are experiencing stress-related complaints originating from work, they will be offered individual work modifications. Conversely, if the issues are unrelated to work, the worker will receive job coaching. As information on this tailored PA approach is lacking, the effectiveness of this approach is investigated. By combining these different intervention components, the investigators strive to fill the research gap concerning the identification of an effective re-integration program for sick-listed workers suffering from stress-related complaints. Participants will be followed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Sick-listed employees from participating organisations (Amsterdam UMC, GGZ inGeest, Rijksschoonmaakorganisatie [RSO], and Transavia)
* Aged 18-68
* Between 2 and 12 weeks on sick leave
* Suffering from stress-related complaints

Exclusion Criteria:

* Non-sick-listed employees
* Suffering from severe psychiatric disorders (e.g., suicidality, mania, psychosis, schizophrenia) or other chronic conditions (e.g., terminal illness) that could significantly affect the employee's mental health and, hence, prevent the return-to work process
* Being pregnant or less than three months after delivery
* Sick-listed for more than 12 weeks
* Inability to complete either the eHealth modules or questionnaires
* Presence of a legal conflict with the employer
* Not signing informed consent

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Lasting return to work | Baseline - 3 months - 6 months -12 months
  Lasting return to work of at least 28 consecutive days without (partial or full) relapse

SECONDARY OUTCOMES:
Stress-related complaints | Baseline - 3 months - 6 months -12 months
  Stress-related complaints (e.g., type of disease, severity of symptoms) by means of the 4DKL (Terluin, 2008), Promis (Terwee et al. 2015).
Psychosocial job characteristics | Baseline - 3 months - 6 months - 12 months
  Psychosocial job characteristics (e.g., mental workload, decision latitude, social support, physical demands, job insecurity) by means of the JCQ (Karasek, Houtman et al. 1995)
Behaviour change | Baseline - 3 months - 6 months - 12 months
  Behaviour change (e.g., attitude, social influence, self-efficacy); by means of the ASE (Damoiseaux et al. 1998), RTW-SE (Volker et al. 2015).

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Amsterdam UMC, Amsterdam
  - GGZ inGeest, Amsterdam
  - Transavia, Amsterdam
  - RSO, The Hague